CLINICAL TRIAL: NCT01249534
Title: Diagnostic Value of C-reactive Protein for Detection of Postoperative Inflammatory Complications After Gastroesophageal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Rene Warschkow, MD, Kantonal Hospital St. Gallen, Department of Visceral Surgery
Other Study IDs: EKSG10/144
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-11

CONDITIONS: Given Indication for Gastroesophageal Cancer Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients after gastroesophageal cancer surgery
  Interventions: Other: gastroesophageal cancer surgery

INTERVENTIONS:
Other: gastroesophageal cancer surgery — gastroesophageal cancer surgery

SUMMARY:
Although widely used, there is a lack of evidence concerning diagnostic value of C-reactive protein (CRP) in the postoperative course. The aim of this study was to evaluate the diagnostic accuracy of CRP for postoperative inflammatory complications after gastroesophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* all patients with gastroesophageal cancer surgery

Exclusion Criteria:

* lack of measurement of C-reactive protein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Given indication for gastroesophageal cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
postoperative Inflammatory complications | 30 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Rene Warschkow, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Department of surgery, Sankt Gallen, Switzerland